CLINICAL TRIAL: NCT02337868
Title: A Double Blind, Randomized, Placebo-Controlled, Phase I Dose Escalation Trial to Evaluate the Safety and Immunogenicity of an Inactivated West Nile Virus Vaccine, HydroVax-001, in Healthy Adults
Brief Title: Phase 1 Trial of Inactivated West Nile Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 13-0020; HHSN272201300017I
Record Dates: First submitted 2015-01-08; First posted 2015-01-14 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2016-12-07

CONDITIONS: West Nile Viral Infection
Keywords: dose-ranging; double blind; female; healthy; HydroVax; male; Placebo-Controlled; Vaccine; West Nile Virus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- High Dose Expanded (Experimental): 15 subjects will receive 4 mcg of HydroVax-001 IM and 4 subjects will receive placebo IM on Days 1 and 29.
  Interventions: Biological: HydroVax-001; Other: Placebo
- High Dose Sentinel (Experimental): 5 subjects will receive 4 mcg of HydroVax-001 IM and 1 subject will receive placebo IM on Days 1 and 29.
  Interventions: Biological: HydroVax-001; Other: Placebo
- Low Dose Expanded (Experimental): 15 subjects will receive 1 mcg of HydroVax-001 IM and 4 subjects will receive placebo IM on Days 1 and 29.
  Interventions: Biological: HydroVax-001; Other: Placebo
- Low Dose Sentinel (Experimental): 5 subjects will receive 1 mcg intramuscularly (IM) of HydroVax-001 and 1 subject will receive placebo IM on Days 1 and 29.
  Interventions: Biological: HydroVax-001; Other: Placebo

INTERVENTIONS:
Biological: HydroVax-001 — HydroVax-001 West Nile Virus inactivated vaccine, alum-adsorbed given at doses of 1 mcg (low dose) and 4 mcg (high dose) IM on days 1 and 29
Other: Placebo — 0.9% Sodium Chloride Injection diluent will be given IM on days 1 and 29

SUMMARY:
This trial will be a randomized, placebo controlled, double-blind (within dosing group), dose escalation phase 1 trial, evaluating dosages of 1 mcg and 4 mcg of HydroVax-001 WNV vaccine given intramuscularly on Day 1 and Day 29 in up to 50 healthy adults > /=18 and < 50 years of age. The primary objective is to assess the safety, reactogenicity, and tolerability of the HydroVax-001 WNV vaccine administered intramuscularly in a two-dose series on Days 1 and 29 at a dose of 1 mcg or a dose of 4 mcg.

DETAILED DESCRIPTION:
This trial will be a randomized, placebo controlled, double-blind (within dosing group), dose escalation phase 1 trial, evaluating dosages of 1 mcg and 4 mcg of HydroVax-001 WNV vaccine given intramuscularly on Day 1 and Day 29 in up to 50 healthy adults > /=18 and < 50 years of age at a single site. The study will consist of two dosing groups of HydroVax-001 vaccine to be enrolled sequentially. Each dose group will consist of 20 individuals who receive HydroVax-001 and 5 who receive placebo. Controls will receive sterile 0.9 percent NaCl placebo intramuscularly at days 1 and 29. The study duration is approximately 25 months (12 month enrollment, 13 month follow up) and subject participation duration of approximately 14 months. The primary objective is to assess the safety, reactogenicity, and tolerability of the HydroVax-001 WNV vaccine administered intramuscularly in a two-dose series on Days 1 and 29 at a dose of 1 mcg or a dose of 4 mcg. The secondary objective is to assess WNV-specific plaque reduction neutralization test (PRNT50) responses after a first dose and after a second dose of HydroVax-001 WNV vaccine given at doses of 1 mcg and 4 mcg. This study aims to recruit up to 50 men and women between the ages of 18 and 50. The study duration is approximately 25 months at a single site and subject participation duration is approximately 14 months.

ELIGIBILITY:
Inclusion Criteria:

1.Age >/=18 years and < 50 years 2.Able to read, sign, and date the informed consent document 3. Available and willing to participate for the planned duration of the study 4.Are in good health, as judged by the investigator and determined by vital signs, medical history, and physical examination 5.Sexually active males must agree to use a medically acceptable form of contraception* in order to be in this study and must agree to continue such use until day 30 after the last vaccination.Medically acceptable contraceptives include: (1) surgical sterilization (such as a vasectomy), or (2) a condom used with a spermicide. Contraceptive measures such as Plan B (TM), sold for emergency use after unprotected sex, are not acceptable methods for routine use. 6.Women of childbearing potential* must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to each vaccination *Not sterilized via tubal ligation, bilateral oophorectomy, or hysterectomy and still menstruating or < 1 year of the last menses if menopausal 7. Women of childbearing potential must have used an acceptable method of contraception* in the 30 days prior to enrollment and must agree to continue such use until day 30 after the last vaccination. *Includes, but is not limited to, abstinence from sex with men,barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing®, successful Essure® placement (permanent, non-surgical, non-hormonal sterilization) with documented confirmation test at least 3 months after the procedure, and licensed hormonal methods such as implants, injectables, or oral contraceptives

Exclusion Criteria:

1. Any clinically significant acute or chronic medical condition* or need for chronic medications** that, in the opinion of the investigator, will interfere with immunity or affect safety *Includes, but is not limited to, disorders of the liver, kidney, lung, heart, or nervous system, or other metabolic or autoimmune/inflammatory conditions ** Receipt of systemic, prescription medications for the treatment of chronic medical conditions or variations of normal physiologic functions are permissible if, in the opinion of the investigator, they are used for conditions that are not clinically significant and would not impact the safety of the subject or the safety and immunogenicity outcomes of the protocol. Use of systemic, over-the-counter medications and PRN systemic, prescription medication are allowed if, in the opinion of the investigator, they pose no additional risk to subject safety or assessment of immunogenicity/reactogenicity. Topical (except corticosteroid) medications, nasal (including corticosteroid) medications, vitamins, and supplements are permissible 2. Asthma, other than mild, well-controlled asthma* *Cold or exercise induced asthma controlled with inhaled medications other than inhaled corticosteroids is permissible. Participants should be excluded if they require daily bronchodilator use, or have had an asthma exacerbation requiring oral/parenteral steroid use or have used theophylline or inhaled corticosteroids in the past year 3. Diabetes mellitus 4. Unstable depression or bipolar disorder* *Has received <3 months of the same anti-depressant or bipolar disorder medication(s) (and dose) or has had a decompensating event during the previous 3 months or has depression or bipolar disorder that in the opinion of the investigator will compromise the subject's ability to comply with protocol requirements 5. Unstable seizure disorder (defined as requiring medication for seizure control or with seizure activity within the past 3 years) 6. Autoimmune disease (lupus, multiple sclerosis, rheumatoid arthritis, autoimmune thyroid disease, etc.); vitiligo, and mild eczema or mild psoriasis not requiring chronic therapy are permissible. 7. Known or suspected congenital or acquired immunodeficiency including anatomic or functional asplenia or immunosupppression as a result of underlying illness or treatment 8. Abuse of alcohol or drugs that, in the opinion of the investigator, may interfere with the subject's ability to comply with the protocol 9. Unstable hypertension (well-controlled hypertension with medication is permissible) 10. Body mass index (BMI) >/= 35 11. Known allergy to components of the study product .Including the following: aluminum hydroxide, sorbitol, potassium chloride, sodium chloride 12. Seropositive to West Nile virus 13. History of a visit to South America or sub-Saharan Africa lasting one month or more 14. History of military service 15. History of vaccination against yellow fever, tick-borne encephalitis, or Japanese encephalitis 16. History of vaccination with West Nile virus candidate vaccines. 17. Attended primary (grade) school in Austria, Germany, Japan, South Korea, India, Thailand, Nepal, Vietnam, or Taiwan (where tick-borne encephalitis vaccine is given) 18. History of dengue fever or receipt of a dengue fever vaccine 19. Active neoplastic disease* *Participants with a history of malignancy may be included if treated by surgical excision or if treated by chemotherapy or radiation therapy has been observed for a period that in the investigator's estimation provides a reasonable assurance of sustained cure (not less than 36 months) 20. Chronic topical or systemic corticoste roid use* *Corticosteroid nasal sprays for allergic rhinitis are permissible. Persons using a topical corticosteroid for a limited duration for mild uncomplicated dermatitis such as poison ivy or contact dermatitis may be enrolled the day after their therapy is completed. Oral or parenteral (intravenous, subcutaneous or intramuscular) corticosteroids given for non-chronic conditions not expected to recur are permissible if, within the year prior to enrollment, the longest course of therapy was no more than 14 days and no oral or parenteral corticosteroids were given within 30 days prior to enrollment. Intraarticular, bursal, tendon, or epidural injections of corticosteroids are permissible if the most recent injection was at least 30 days prior to enrollment. 21. Are breastfeeding or plan to breastfeed at any time throughout the study 22. Receipt or planned receipt of inactivated vaccine or allergy desensitization injection 14 days before or after a study vaccination 23. Receipt or planned receipt of live attenuated vaccine 30 days before or after a study vaccination 24. Receipt of any other experimental agent within 30 days prior to vaccination or planned receipt prior to the end of the study 25. Plans to enroll in another clinical trial* that could interfere with safety assessment of the investigational product at any time during the study period *Includes trials that have a study intervention such as a drug, biologic, or device 26 Receipt of blood products or immunoglobulin within six months prior enrollment 27. Donation of a unit of blood within 56 days prior to enrollment or intends to donate blood during the study period 28. Systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg 29.Resting heart rate <40 or >100 beats per minute 30.Oral temperature >/= 38 degrees C (100.4 degrees F) 31.Positive serology for HIV 1/2* *If the enzyme linked immunosorbent assay (ELISA) is positive, HIV confirmation should be performed. If the HIV Western Blot is not consistent with HIV infection, the volunteer may be enrolled. A past participant in an HIV vaccine trial who has a positive antibody ELISA may participate if the Western Blot is not consistent with pending seroconversion or positive or an HIV polymerase chain reaction (PCR) assay result is below the level of detection of HIV. 32. Positive hepatitis B surface antigen (HBsAg) 33. Positive antibody to hepatitis C virus (HCV) 34. Any Grade 1 or higher screening clinical lab value* (see Toxicity Table Appendix B) *Screening clinical labs include blood tests (white blood cell [WBC] count, hemoglobin level, platelet count, creatinine, blood urea nitrogen, non-fasting glucose, potassium, alanine aminotransferase [ALT], aspartate aminotransferase [AST], and total bilirubin) and urine tests (protein, glucose). 35. Plan to have a major change in exercise routine from 72 hours before any dose of study vaccine/placebo through 15 days after that dose 36. Acute febrile illness (oral temperature >/= 38 deg

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Occurrence of any AE related to the study vaccine through day 57 after the second vaccination | Day 1 post first vaccination to Day 57 post second vaccination
Occurrence of Grade 3 laboratory toxicities related to the study vaccine from first vaccination through day 15 after the second vaccination | Day 1 post first vaccination to Day 15 post second vaccination
Occurrence of Grade 3 unsolicited adverse events related to the study vaccine from first vaccination through day 57 after the second vaccination | Day 1 post first vaccination to Day 57 post second vaccination
Occurrence of SAEs related to the study vaccine at any time during the study | Day 1 post first vaccination to Day 365 post second vaccination
Occurrence of solicited local AE and reactogenicity signs and symptoms in the 14 days after each vaccination | Day 1 post first vaccination to Day 14 post first and second vaccination
Occurrence of solicited systemic AE and reactogenicity signs and symptoms in the 14 days after each vaccination | Day 1 post first vaccination to Day 14 post first and second vaccination

SECONDARY OUTCOMES:
Geometric mean PRNT50 titer at days 15 and 29 after first vaccination and at days 15, 29, 57, 180, and 365 following second vaccination | Days 15 and 29 post first vaccination and Days 15, 29, 57, 180, and 365 post second vaccination
Percentage of subjects achieving seroconversion in PRNT50 titer (fourfold or greater increase in titer from baseline) at day 29 after first vaccination and at day 57 after second vaccination | Day 29 post first vaccination and Day 57 post second vaccination
The reverse cumulative distribution curve of PRNT50 titer on Days 15 and 29 after first vaccination and at days 15, 29, 57, 180, and 365 after the second vaccination for each dose group and for all dose groups combined | Days 15 and 29 post first vaccination and Days 15, 29, 57, 180, and 365 post second vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Human Vaccine Institute - Duke Clinical Vaccine Unit, Durham, North Carolina, United States